CLINICAL TRIAL: NCT05758285
Title: Using Responsible Artificial Intelligence (AI) to Predict Online Therapy Outcome and Engagement
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02263; th23Meinlschmidt
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Mental Health Care; Mental Disorders
Keywords: Artificial Intelligence (AI); Digital Therapeutics (DTx); Internet-delivered, Cognitive Behaviour Therapy (iCBT); Information and Communication Technology (ICT); Explainable Artificial Intelligence (XAI); Digital psychotherapy; Personalised prediction models; Bias; AI-based prediction models; Online Therapy Unit; Anxiety symptoms; Depressive symptoms; Wellbeing Course
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders; Depression | interventions — Treatment Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AI-Based Prediction of Treatment Engagement and Outcomes — AI-based algorithms and prediction models of treatment engagement and outcomes based on data from the Online Therapy Unit by Prof. Heather Hadjistavropoulos will be trained to predict symptom improvement of patients from pre- to post-digital psychotherapy intervention and to predict patients' engagement with the digital psychotherapy intervention and to predict patient drop out probability. For prediction model estimation, state of the art AI-based algorithms, such as XGBoost, is used . XGBoost is a machine learning method developed by refining previously established decision-tree-based methodologies. Data is split into training and testing sets (e.g., 80/20 split).

SUMMARY:
This study is to develop AI-based models for the personalised prediction of treatment engagement and treatment outcomes in patients engaging in digital psychotherapy. A large, real-world dataset of patients in a digital psychotherapy program will be used to train AI algorithms. Responsible AI algorithms will be developed by describing, accounting for, and mitigating bias due to severity of mental disturbances in AI-based models, in addition to considering bias due to other sensitive attributes, such as gender, ethnicity, and socio-demographic status.

DETAILED DESCRIPTION:
Mental disorders contribute greatly to the global disease burden, but many people do not have access to mental health care. This treatment gap is partly due to structural (e.g., availability) and attitude-related (e.g. fear of stigma) barriers in health care seeking. Digital therapeutics (DTx) in the form of digital mental health interventions or digital psychotherapy may be the solution to this problem. The integration of Information and Communication Technology (ICT) and mental health care has the potential to increase the efficiency of care delivery and enables personalisation of treatments. Artificial Intelligence (AI)-based analysis of large datasets from digital psychotherapy programs may allow developing and validating personalised prediction models. The prediction of individual engagement and the early identification of untoward engagement patterns may improve personalisation of DTx, which could help reduce nonadherence and improve treatment outcome. The personalised prediction of DTx outcomes and engagement patterns may be achieved by implementing AI-based approaches, such as Machine Learning prediction models. Personalised prediction models may lead to a better understanding of who profits most from what kind of DTx in a real-world setting. Taken together, personalisation of DTx treatment outcomes and engagement may i) improve decision making processes in patient-clinician dyads, ii) improve efficiency of digital psychotherapy, iii) reduce suffering of patients, and iv) reduce direct and indirect cost related to mental health care. There is a need to account for potential discrimination due to mental health in AI-based predictions models. Unbiased and non- discriminating AI is often referred to as responsible AI. Accounting for bias in AI-based prediction models based on a specific dataset is especially important in mental health care to prevent acceleration of health discrimination.

This study is to develop AI-based models for the personalised prediction of treatment engagement and treatment outcomes in patients engaging in digital psychotherapy. A large, real-world dataset of patients in a digital psychotherapy program will be used to train AI algorithms. Responsible AI algorithms will be developed by describing, accounting for, and mitigating bias due to severity of mental disturbances in AI-based models, in addition to considering bias due to other sensitive attributes, such as gender, ethnicity, and socio-demographic status. The aim of the proposed project is to estimate AI-based prediction models of treatment engagement and outcomes based on data from the Online Therapy Unit by Prof. Heather Hadjistavropoulos from the University of Regina, Canada. The Online Therapy Unit dataset contains a large amount of data on DTx from people with mental disorders (collected as part of research trials in the Online Therapy Unit from 2013 to 2021) and is derived from the publicly funded, internet-delivered, cognitive behaviour therapy (iCBT) program in Saskatchewan, Canada. In sum, the Online Therapy Unit dataset is highly suitable as a training and test dataset for AI-based prediction models, as it comprises a large number of participants, longitudinal data retrieved from the real world opposed to a clinical trial, and a rich set of predictive features.

ELIGIBILITY:
Inclusion Criteria:

* Participants that were screened as eligible to take part in a Wellbeing Course trial offered at the Online Therapy Unit between Nov 4 2013 and Dec 21 2021.
* Participants that consented to the use of their data to evaluate and improve iCBT services.
* Accessed Lesson 1 of the course content and completed baseline questionnaires.

Exclusion Criteria:

* Data will only be excluded in case of errors in data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants at the publicly funded, internet-delivered, cognitive behaviour therapy (iCBT) program in Saskatchewan, Canada. The program provides symptom screenings and an eight-week transdiagnostic iCBT program called the Wellbeing Course. In Saskatchewan, this transdiagnostic iCBT program has been integrated into the public mental health care, for example by assigning clinicians in community mental health clinics to the Online Therapy Unit and by encouraging therapists to direct patients to this service. Data was collected as part of research trials in the Online Therapy Unit from 2013 to 2021.
Sampling Method: Probability Sample
Enrollment: 6671 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire 9-item (PHQ9) (percent change) | week 1 until week 8
  Change in PHQ9 (percent change) to evaluate symptom improvement vs. no symptom improvement pre- to post-digital psychotherapy intervention. Patient Health Questionnaire (PHQ-9): Total = /27 ; Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Change in General Anxiety Disorder-7 Questionnaire (GAD7) (percent change) | week 1 until week 8
  Change in General Anxiety Disorder-7 Questionnaire (GAD7) to evaluate symptom improvement vs. no symptom improvement pre- to post-digital psychotherapy intervention. Score 0-4: Minimal Anxiety · Score 5-9: Mild Anxiety · Score 10-14: Moderate Anxiety · Score greater than 15: Severe Anxiety.

OTHER OUTCOMES:
Number of messages sent by client | week 1 until week 8
  Patients' engagement with the digital psychotherapy intervention by assessing the number of patient messages
Number of messages received by client | week 1 until week 8
  Patients' engagement with the digital psychotherapy intervention by assessing the number of therapist messages
Number of phone calls to physician notes | week 1 until week 8
  Patients' engagement with the digital psychotherapy intervention by assessing the number of phone calls
Number of times client logged in | week 1 until week 8
  Patients' engagement with the digital psychotherapy intervention by assessing the number of lessons accessed

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Prof., Principal Investigator — University Hospital Basel, Department of Psychosomatic Medicine
Locations (1):
- University Hospital Basel, Department of Psychosomatic Medicine, Basel, Switzerland

REFERENCES:
- [Result] Roemmel N, Bahmane S, Hadjistavropoulos HD, Nugent M, Lieb R, Meinlschmidt G. Prediction of treatment outcome in patients receiving internet-delivered cognitive behavioural therapy for depressive and anxiety symptoms: a machine learning analysis of data from a healthcare-embedded longitudinal study. BMJ Open. 2025 Sep 3;15(9):e097651. doi: 10.1136/bmjopen-2024-097651. PMID 40903086